CLINICAL TRIAL: NCT07149909
Title: The Clinical Effect of Fiberoptic Bronchoscopy in Management of Adult Patients With Severe Ventilator-associated Pneumonia; a Randomized Controlled Trial
Brief Title: Fiberoptic Bronchoscopy in Severe Ventilator-associated Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Gehad Mohamed Mohsen Mahmoud, Assistant Lecturer of Critical Care Medicine, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD: 8-11-2023
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Ventilator-Associated Pneumonia; Severe Pneumonia; Critical Illness
Keywords: Fiberoptic bronchoscopy; Bronchoalveolar lavage (BAL); Mechanical ventilation; Intensive care unit (ICU); Respiratory infection; Secretion clearance; Culture-directed antibiotics; Severe VAP
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pneumonia; Critical Illness; Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to receive either standard therapy alone or standard therapy plus fiberoptic bronchoscopy.
Masking Description: This was an open-label trial; neither participants, care providers, nor investigators were blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants received standard therapy for severe ventilator-associated pneumonia, which included culture-guided antibiotics, routine drug therapy, tracheal lavage, and aspiration. Sputum samples were collected for bacterial culture and sensitivity testing to guide antibiotic selection.
  Interventions: Other: Other (Conventional Therapy)
- Fiberoptic Bronchoscopy Group (Experimental): Participants received the same standard therapy as the control group plus fiberoptic bronchoscopy. The bronchoscope was inserted via the endotracheal tube to clear secretions, obtain samples for culture, and perform bronchoscopic alveolar lavage. Lavage was performed once daily for one week using sterile sodium chloride solution with ambroxol hydrochloride, followed by antibiotic administration. Cultures were used to guide therapy.
  Interventions: Procedure: Fiberoptic Bronchoscopy

INTERVENTIONS:
Other: Other (Conventional Therapy) — Participants received standard therapy including culture-guided antibiotics, tracheal lavage, and aspiration. Sputum samples were collected from the lower trachea for culture and sensitivity testing to guide antibiotic selection.
  Arms: Control Group
Procedure: Fiberoptic Bronchoscopy — Participants underwent fiberoptic bronchoscopy through the endotracheal tube for secretion clearance, sample collection, and alveolar lavage once daily for one week. Sterile sodium chloride solution with ambroxol hydrochloride was instilled, and antibiotics were administered immediately after lavage. Samples were cultured to guide antibiotic therapy.
  Arms: Fiberoptic Bronchoscopy Group

SUMMARY:
This randomized controlled trial evaluated the clinical effect of fiberoptic bronchoscopy in the management of adult patients with severe ventilator-associated pneumonia (VAP). A total of 100 patients admitted to the Critical Care Department at Benha University Hospitals were enrolled and randomly assigned in equal numbers to two groups. The control group received standard therapy, including culture-guided antibiotics, lavage, and aspiration. The intervention group received the same treatment plus fiberoptic bronchoscopy for secretion clearance, lavage, and culture-directed antibiotic therapy.

The primary outcome was the overall effective treatment rate, defined as the proportion of patients with significant or partial clinical improvement. Secondary outcomes included recovery time, length of intensive care unit stay, respiratory mechanics, inflammatory markers (C-reactive protein and procalcitonin), recurrence of pulmonary infection, and 28-day mortality.

The study demonstrated whether the addition of fiberoptic bronchoscopy to conventional treatment improved clinical outcomes in patients with severe ventilator-associated pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Patients of both sexes
* Patients requiring mechanical ventilation
* Development of pneumonia ≥ 48 hours after endotracheal intubation or ≥ 48 hours after extubation
* Diagnosis of severe ventilator-associated pneumonia defined by a Modified Clinical Pulmonary Infection Score (CPIS) > 6

Exclusion Criteria:

* Refusal to participate
* Presence of lung shadows prior to mechanical ventilation
* Severe bleeding disorders or immune system diseases
* Severe hemodynamic instability
* Recent myocardial infarction or unstable arrhythmia
* Tracheal stenosis or upper airway mass

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Overall Effective Treatment Rate | Postoperatively (within 28 days of VAP diagnosis).
  Proportion of patients achieving significant or partial clinical improvement based on resolution of symptoms, normalization of temperature and laboratory markers, negative sputum cultures, and radiologic improvement.

SECONDARY OUTCOMES:
Recovery Time | Up to 28 days from diagnosis.
  Duration from diagnosis of ventilator-associated pneumonia (VAP) until Modified Clinical Pulmonary Infection Score (CPIS) decreased to below 6.
Length of intensive care unit (ICU) stay | From intensive care unit (ICU) admission until discharge (maximum 28 days).
  Total number of days spent in the intensive care unit during the hospital admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, Benha, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (de-identified) that underlie the results reported in this trial will be made available to qualified researchers upon reasonable request for the purpose of meta-analyses and further research on ventilator-associated pneumonia management.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: De-identified individual participant data and supporting documents will be available beginning 6 months after publication of the main study results and for up to 5 years thereafter.
Access Criteria: Researchers who provide a methodologically sound proposal will be granted access after review and approval by the principal investigator and the Research Ethics Committee of Benha Faculty of Medicine. Data will be shared through secure data transfer agreements to ensure confidentiality.